CLINICAL TRIAL: NCT04287790
Title: Promoting Medications for Alcohol Use Disorder on the General Medicine Service at Yale New Haven Hospital: a Pilot Study
Brief Title: Promoting Medications for Alcohol Use Disorder on the General Medicine Service
Status: Terminated | Type: Observational
Why Stopped: COVID-19 disrupted recruitment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000026722
Record Dates: First submitted 2020-02-17; First posted 2020-02-27 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Use Disorder
Keywords: Implementation; Medications for alcohol use disorder; Pharmacotherapy
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate; Naltrexone; Disulfiram; Ethanol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Health professionals after intervention: Health professionals (physicians, advanced practice providers, pharmacists, social workers, and nurses) who work on the designated general medicine services at Yale New Haven Hospital after implementation intervention (July 2020)
  Interventions: Behavioral: audit and feedback, educational meetings, and academic detailing to promote medication receipt
- Hospitalized patient before intervention: Patients discharged from the general medicine service at Yale New Haven Hospital York street campus following hospitalization for an alcohol related diagnosis 18 months before the start (January 1st 2020) of the implementation intervention
  Interventions: Drug: Acamprosate, naltrexone, or disulfiram
- Health professionals before intervention: Health professionals (physicians, advanced practice providers, pharmacists, social workers, and nurses) who work on the designated general medicine services at Yale New Haven Hospital after implementation intervention (December 2019)
- Hospitalized patient after intervention: Patients discharged from the general medicine service at Yale New Haven Hospital York street campus following hospitalization for an alcohol related diagnosis 12 months after the start (January 1st 2020) of the implementation intervention
  Interventions: Drug: Acamprosate, naltrexone, or disulfiram

INTERVENTIONS:
Behavioral: audit and feedback, educational meetings, and academic detailing to promote medication receipt — Our implementation intervention will incorporate the following strategies: 1) Formation of an alcohol-related care working group. This voluntary working group will consist of members of the research team and volunteer health professionals from YNHH. The group with supervise and support the other intervention components. 2) We will develop medication for alcohol use disorder marketing (posters and buttons) materials and educational (pamphlet) materials and distribute these materials to health professionals. 3) Building on the existing infrastructure and collaboration, the research team will assist in revising existing alcohol-related care daily monitoring systems to support auditing and feedback on the adoption of medications for alcohol use disorder at YNHH. 4) The research team will hold educational meetings and educational outreach visits (academic detailing) when invited during regular noon conferences and team meetings.
  Groups: Health professionals after intervention
Drug: Acamprosate, naltrexone, or disulfiram — Increased receipt of medications for alcohol use disorder facilitated by the implementation intervention.
  Other Names: FDA medications for alcohol use disorder
  Groups: Hospitalized patient after intervention; Hospitalized patient before intervention

SUMMARY:
Medications for Alcohol use disorder (MAUD) (acamprosate, naltrexone, and disulfiram) remain underutilized despite guideline recommendations and rising alcohol-related morbidity and mortality. Alcohol use disorder (AUD)-related hospitalizations are opportunities to initiate MAUD, but optimal implementation strategies are unclear. We will complete a 6 month pilot implementation intervention involving audit and feedback, educational meetings, and academic detailing for health professionals at Yale New Haven Hospital to determine the impact on: 1) health professional satisfaction with intervention components, 2) health professional knowledge and attitudes about medications for alcohol use disorder, 3) receipt of medication among hospitalized patients diagnosed with an alcohol use disorder and 4) 30 day readmission among hospitalized patients with alcohol use disorder. Health professional satisfaction and knowledge with be assessed using a pre-post design and receipt of medications and 30 day readmission will be assessed using a interrupted time series design. We hypothesize health professional knowledge and attitudes about MAUD will be greater after the pilot intervention compared to before. We hypothesize receipt of MAUD will be greater after the pilot intervention compared to before. We hypothesize 30 day readmission will be less after the pilot intervention compared to before.

DETAILED DESCRIPTION:
Medications for Alcohol use disorder (MAUD) (acamprosate, naltrexone, and disulfiram) remain underutilized despite guideline recommendations and rising alcohol-related morbidity and mortality. Alcohol use disorder (AUD)-related hospitalizations are opportunities to initiate MAUD, but optimal implementation strategies are unclear. We will complete a 6 month pilot implementation intervention involving audit and feedback, educational meetings, and academic detailing for health professionals at Yale New Haven Hospital (YNHH) to determine the impact on: 1) health professional satisfaction with intervention components, 2) health professional knowledge and attitudes about medications for alcohol use disorder, 3) receipt of medication among hospitalized patients diagnosed with an alcohol use disorder and 4) 30 day readmission among hospitalized patients with alcohol use disorder. Health professional satisfaction and knowledge with be assessed using a pre-post design and receipt of medications and 30 day readmission will be assessed using a interrupted time series design. We hypothesize health professional knowledge and attitudes of MAUD will be greater after the pilot intervention compared to before. We hypothesize receipt of MAUD will be greater after the pilot intervention compared to before. We hypothesize 30 day readmission will be less after the pilot intervention compared to before.

Population and setting for implementation intervention:

Health professionals (physicians, advanced practice providers, pharmacists, social workers, and nurses) who work on the designated general medicine services (9-5, 4-6 and 4-7) at Yale New Haven Hospital.

Implementation intervention:

Our implementation intervention will incorporate the following strategies: 1) Formation of an alcohol-related care working group. This voluntary working group will consist of members of the research team and volunteer health professionals from YNHH. The group with supervise and support the other intervention components. 2) We will develop medication for alcohol use disorder marketing (posters and buttons) materials and educational (pamphlet) materials and distribute these materials to health professionals. 3) Building on the existing infrastructure and collaboration, the research team will assist in revising existing alcohol-related care daily monitoring systems to support auditing and feedback on the adoption of medications for alcohol use disorder at YNHH. 4) The research team will hold educational meetings and educational outreach visits (academic detailing) when invited during regular noon conferences and team meetings.

Health professional outcomes: health professional satisfaction and knowledge Using the pre-post design, data collection will consist of two surveys. One survey will assess health professional knowledge and attitudes about MAUD at baseline and then again at 6 months post intervention. A follow up survey will assess health professional satisfaction with the intervention components collected following educational events and at 6 months post intervention.

Patients with AUD outcomes: receipt of medication among hospitalized patients diagnosed with an alcohol use disorder (primary outcome) and 30 day readmission among patient with alcohol use disorder. Using an interrupted time series design, data will be obtained from Epic electronic medical record at Yale New Haven Hospital in partnership with the Joint Data Analytics Team (JDAT) to whom we will submit our formal data request. Patients discharged from the general medicine service at Yale New Haven Hospital York street campus following hospitalization for an alcohol related diagnosis 18 months before and 12 months after the start (January 1st 2020) of the implementation intervention.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals (physicians, advanced practice providers, pharmacists, social workers, and nurses) who work on the 9-5, 4-6 and 4-7 general medicine services at Yale New Haven Hospital. The intervention will be conducted on 9-5, 4-6 and 4-7 general medicine services at Yale New Haven Hospital.

Exclusion Criteria:

* Physicians trainees (student, residents, and fellows) will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Health professionals (physicians, advanced practice providers, pharmacists, social workers, and nurses) who work on the 9-5, 4-6 and 4-7 general medicine services at Yale New Haven Hospital. The intervention will be conducted on 9-5, 4-6 and 4-7 general medicine services at Yale New Haven Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Before and after intervention change in receipt of medication | 18 months before and 12 months after the start (January 1st 2020) of the implementation intervention
  receipt of medication among hospitalized patients diagnosed with an alcohol use disorder (patients discharged from the general medicine service at Yale New Haven Hospital York street campus following hospitalization for an alcohol related diagnosis) The primary outcome, receipt of medication, can occur with any of four events:
  1. Administration of intramuscular naltrexone during hospitalization (Y/N)
  2. Discharge outpatient prescription of acamprosate (Y/N)
  3. Discharge outpatient prescription of naltrexone (Y/N)
  4. Discharge outpatient prescription of disulfiram (Y/N)

SECONDARY OUTCOMES:
Before and after intervention change in 30 day readmission | 18 months before and 12 months after the start (January 1st 2020) of the implementation intervention
  30 day readmission (Y/N) among hospitalized patients with alcohol use disorder. Patients discharged from the general medicine service at Yale New Haven Hospital York street campus following hospitalization for an alcohol related diagnosis
Before and after intervention change in health professional acceptability | December 2019 and July 2020
  Pre-post Acceptability Rating Profile survey, maximum value 6 and minimum value 1 with higher scores indicating greater acceptability
Before and after intervention change in health professional knowledge | December 2019 and July 2020
  Pre-post survey adapted Physician Competence in Substance Abuse Test
Before and after intervention change in health professional appropriateness | December 2019 and July 2020
  Pre-post Parenting Strategies Questionnaire, maximum 6 and minimum 1 with higher scores indicating greater appropriateness
Before and after intervention change in health professional feasibility | December 2019 and July 2020
  Pre-post Ratings of Threshold Assessment Grid feasibility, maximum 6 and minimum 1 with higher scores indicating greater feasibility
Post intervention acceptability of education materials among health professionals | July 2020
  Post intervention Manual Acceptability Rating Scale, maximum 3 and minimum 1 with higher scored indicating great acceptability of educational materials

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Joudrey, MD MPH, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No